CLINICAL TRIAL: NCT00550693
Title: A Crossover Intervention Trial Evaluating the Efficacy of a Chlorhexidine-Impregnated Sponge (BIOPATCH®) to Reduce Catheter-Related Bloodstream Infections in Hemodialysis Patients
Brief Title: Trial Evaluating the Efficacy of a Chlorhexidine-Impregnated Sponge (BIOPATCH®) to Reduce Catheter-Related Bloodstream Infections in Hemodialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Biopatch 400-05-005; WUSM HRPO 04-1312
Record Dates: First submitted 2007-10-29; First posted 2007-10-30 (Estimated); Last update posted 2007-10-30 (Estimated); Status verified 2007-10

CONDITIONS: Catheter Related Bloodstream Infection
Keywords: bloodstream infections; hemodialysis catheter
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Placebo Comparator): The patients in this arm continued with the local catheter care protocol.
  Interventions: Device: Chlorhexidine-impregnated foam dressing

INTERVENTIONS:
Device: Chlorhexidine-impregnated foam dressing — Patients during the intervention period had this foam dressing applied around their central venous catheter. This was replaced once a week as recommended by the package insert unless the dressing was soiled, bloody, or fell off.
  Other Names: Biopatch Antimicrobial Dressing

SUMMARY:
There are currently no published data on the efficacy of the chlorhexidine-impregnated foam dressing to reduce catheter-related bloodstream infections (BSI) in hemodialysis patients.

The researchers perfomed a cross-over intervention trial on patients who were dialyzed through central venous catheters at two outpatient dialysis centers were enrolled. The use of a chlorhexidine-impregnated foam dressing was incorporated into the catheter care protocol during the intervention period. A nested cohort study of all patients who received the foam dressing was also conducted to determine independent risk factors for development of BSI.

The primary outcomes were the catheter-related bloodstream infection rates in the intervention and control groups. Secondary outcomes include the clinical sepsis rates between the two groups and risk factors for development of bloodstream infection despite the use of the foam dressing.

ELIGIBILITY:
Inclusion Criteria:

* All patients who were dialyzed through a central venous catheter during the time period

Exclusion Criteria:

* Patients who were allergic to chlorhexidine

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2004-04; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Catheter-related bloodstream infection rate in bloodstream infections/1000 dialysis sessions | over a six-month period

SECONDARY OUTCOMES:
clinical sepsis rates between the two groups; exit site infection rates between the two groups; adverse events related to the intervention | over a 6 month period

CONTACTS AND LOCATIONS:
Overall Officials: Bernard C Camins, MD, MSCR, Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - Barnes-Jewish Dialysis Center, St Louis, Missouri
  - Chromalloy American Kidney Center, St Louis, Missouri